CLINICAL TRIAL: NCT00945984
Title: Comparison of Laparoendoscopic Single-site Radical Nephrectomy With Conventional Laparoscopic Radical Nephrectomy for Localized Renal Cell Carcinoma
Brief Title: Laparoendoscopic Single-site Radical Nephrectomy for Localized Renal Cell Carcinoma
Acronym: LESS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hyeon Hoe Kim, Seoul National University Hospital
Other Study IDs: LESSRNx
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Localized Renal Cell Carcinoma
Keywords: Localized renal cell carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- LESS: Patients who underwent LESS radical nephrectomy
  Interventions: Procedure: Radical nephrectomy
- Conventional laparoscopy: Patients who underwent conventional laparoscopic radical nephrectomy
  Interventions: Procedure: Radical nephrectomy

INTERVENTIONS:
Procedure: Radical nephrectomy — Surgical options to treat localized renal cell carcinoma

SUMMARY:
Surgical resection is the only potential curative treatment available for renal cell carcinoma. The purpose of this study is to clarify the surgical and oncologic outcomes of laparoendoscopic single-site radical nephrectomy for localized Renal Cell Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized renal cell carcinoma

Exclusion Criteria:

* Patients with lymph node or distant metastasis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary care center
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-03

PRIMARY OUTCOMES:
Surgical outcomes such as operative time, estimated blood loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon Hoe Kim, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea